CLINICAL TRIAL: NCT00532155
Title: A Multinational, Randomized, Double-Blind Study Comparing Aflibercept Versus Placebo in Patients Treated With Second-Line Docetaxel After Failure of One Platinum Based Therapy for Locally Advanced or Metastatic Non-Small-Cell Lung Cancer
Brief Title: A Study of Aflibercept Versus Placebo in Patients With Second-Line Docetaxel for Locally Advanced or Metastatic Non-Small-Cell Lung Cancer
Acronym: VITAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC10261; EudraCT 2007-000819-29
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma; Non Small Cell Lung
Keywords: lung cancer; angiogenesis inhibitor; chemotherapy
MeSH Terms: conditions — Carcinoma; Lung Neoplasms | interventions — aflibercept; Docetaxel; Dexamethasone; Lead

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aflibercept/Docetaxel (Experimental): Participants with Non-Small-Cell Lung Cancer (NSCLC) were administered Aflibercept immediately followed by Docetaxel every three weeks until disease progression, unacceptable toxicity, or participant's refusal.
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®); Drug: Docetaxel (Taxotere®); Drug: Dexamethasone (pre- and post-medication for docetaxel)
- Placebo/Docetaxel (Placebo Comparator): Participants with Non-Small-Cell Lung Cancer (NSCLC) were administered Placebo immediately followed by Docetaxel every three weeks until disease progression, unacceptable toxicity, or participant's refusal.
  Interventions: Drug: Placebo; Drug: Docetaxel (Taxotere®); Drug: Dexamethasone (pre- and post-medication for docetaxel)

INTERVENTIONS:
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 6 mg/kg Aflibercept administered intravenously (IV) over 1 hour once on Day 1, every 3 weeks.
  Arms: Aflibercept/Docetaxel
Drug: Placebo — Matching placebo to Aflibercept administered intravenously (IV) over 1 hour once on Day 1, every 3 weeks.
  Arms: Placebo/Docetaxel
Drug: Docetaxel (Taxotere®) — 75 mg/m² docetaxel in 250 mL dextrose 5% or NaCl 0.9% administered intravenously (IV) over 1 hour, on Day 1 every 3 weeks.
Drug: Dexamethasone (pre- and post-medication for docetaxel) — As a pre- and post-medication for docetaxel, 8 mg dexamethasone was administered orally, the evening before Day 1, on Day 1 (early morning, 1 hour before docetaxel treatment, and evening) and on Day 2 (morning and evening).

SUMMARY:
The primary objective of the study was to demonstrate overall survival improvement for aflibercept + docetaxel compared to docetaxel + placebo as second line treatment for participants with locally advanced or metastatic non-small cell lung cancer (NSCLC).

The secondary objectives were to compare other efficacy parameters, to assess the overall safety of the two treatment arms, to assess the pharmacokinetics of intravenous (IV) aflibercept in this participant population and to determine immunogenicity of IV aflibercept in all participants.

DETAILED DESCRIPTION:
The study included:

* A screening visit of up to 21 days prior to randomization
* Randomization at baseline (Treatment was initiated with 3 days of randomization)
* A treatment period with 3-week treatment cycles until the participant met the following discontinuation criteria: had progressive disease, had unacceptable toxicity, or refused further study treatment
* A post study treatment follow-up period (a visit was scheduled every 8 weeks until death or end of study)

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological proven locally advanced or metastatic non-small cell lung cancer
* Disease progression during or after one, and only one, prior anticancer therapy which is platinum-based for advanced or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Adequate renal, liver and bone marrow functions

Exclusion Criteria:

* Squamous histology/cytology
* Less than 28 days elapsed from prior treatment with radiotherapy, surgery, or chemotherapy to the time of randomization
* Prior isotope therapy, whole pelvic radiotherapy, or radiotherapy to > 25% of bone marrow
* Prior docetaxel treatment
* Uncontrolled hypertension

The above information was not intended to contain all considerations relevant to participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administraive Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Admnistrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Ramlau R, Gorbunova V, Ciuleanu TE, Novello S, Ozguroglu M, Goksel T, Baldotto C, Bennouna J, Shepherd FA, Le-Guennec S, Rey A, Miller V, Thatcher N, Scagliotti G. Aflibercept and Docetaxel versus Docetaxel alone after platinum failure in patients with advanced or metastatic non-small-cell lung cancer: a randomized, controlled phase III trial. J Clin Oncol. 2012 Oct 10;30(29):3640-7. doi: 10.1200/JCO.2012.42.6932. Epub 2012 Sep 10. PMID 22965962

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1130 participants signed an informed consent to enter the study. Amongst these, 913 were randomized to the two arms in this study. 217 participants were screen failures.
Period: Overall Study
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Started | 457 | 456
SAFETY POPULATION | 455 | 450
Completed | 0 (Participants continued treatment until they met treatment discontinuation criteria) | 0 (Participants continued treatment until they met treatment discontinuation criteria)
Not Completed | 457 | 456
Not completed — Adverse Event | 66 | 123
Not completed — Lack of Efficacy | 332 | 255
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 16 | 15
Not completed — Withdrawal by Subject | 23 | 44
Not completed — Consent withdrawn | 5 | 7
Not completed — Moved | 1 | 0
Not completed — Pre-existing brain metastasis (by MRI) | 1 | 0
Not completed — Occurence of a second cancer | 0 | 1
Not completed — Occurence of a secondary cancer | 0 | 1
Not completed — Promotor ended study | 1 | 0
Not completed — Progressive disease (by incorrect scan) | 0 | 1
Not completed — Had brain metastasis, was mis-randomized | 1 | 0
Not completed — Study stopped | 1 | 0
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Study termination stop further treatment | 4 | 0
Not completed — Did not receive study medication | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel | Total
Number analyzed (Participants) | 457 | 456 | 913
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (9.4) | 59.6 (9.5) | 59.6 (9.4)
Age, Customized [Number; unit: participants]
  <65 years | 316 | 315 | 631
  >= and <75 years | 122 | 121 | 243
  >=75 years | 19 | 20 | 39
Sex/Gender, Customized [Number; unit: participants]
  Male | 300 | 305 | 605
  Female | 157 | 151 | 308
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 405 | 411 | 816
  Black | 10 | 7 | 17
  Asian/Oriental | 40 | 34 | 74
  Other | 2 | 4 | 6
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.8 (0.2) | 1.8 (0.2) | 1.8 (0.2)
Prior Bevacizumab (as per IVRS) [Number; unit: participants] — Number of participants who had received prior bevacizumab as per interactive voice response system (IVRS).
  participants
    Yes | 53 | 51 | 104
    No | 404 | 405 | 809
Eastern Cooperative Oncology Group (ECOG) performance status score (as per IVRS) [Number; unit: participants] — The ECOG score assesses how the disease affects a participant's daily living abilities. It ranges from 0-5, with 0 being the best and 5 being the worst outcome. "0" reflects a fully active participant, able to carry on all pre-disease performance without restriction. "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. "2" reflects an ambulatory participant, who is up and about more than 50% of waking hours, and capable of all self-care but unable to carry out any work activities.
  participants
    Participants with ECOG Score = 0 | 151 | 149 | 300
    Participants with ECOG Score = 1 | 283 | 286 | 569
    Participants with ECOG Score = 2 | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was time interval from the date of randomization to the date of death due to any cause. If death was not observed during the study, overall survival time was censored at the last date the participant was known to be alive, or the study cutoff date, whichever was earlier. The cut-off date for the OS was date when 687 deaths were observed.
  OS was estimated from Kaplan-Meier Curves.
Time Frame: Baseline to the date when 687 deaths occurred (26 January 2011)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Events (Death)
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Number analyzed (Participants) | 457 | 456
Number analyzed (Events (Death)) | 344 | 343
months | 10.41 [9.199 to 11.860] | 10.05 [9.166 to 11.598]
Statistical Analysis 1: Comparison: Placebo/Docetaxel vs Aflibercept/Docetaxel; Test type: Superiority or Other; p = 0.8985, Stratified log-rank test; Stratified on ECOG Performance Status (0 vs 1 vs 2) and Prior Bevacizumab (yes vs no) according to IVRS; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.868 to 1.174]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval between the date of randomization and the time of occurrence of the first radiological tumor progression detected by a computer tomography (CT) scan and /or by Magnetic Resonance Imaging (MRI); or death due to any cause; whichever was earlier. Participants without disease progression were censored at the earliest date between their last valid tumour assessment and the data cutoff date.
  PFS was estimated from Kaplan-Meier Curves.
Time Frame: Baseline to data cut-off (26 January 2011)
Population: Intent to treat (ITT) population. The results are based on a total of 865 PFS events (434 in the placebo group and 431 in the aflibercept group) at the time of cutoff.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: PFS Events
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Number analyzed (Participants) | 457 | 456
Number analyzed (PFS Events) | 434 | 431
months | 4.11 [3.515 to 4.337] | 5.19 [4.370 to 5.552]
Statistical Analysis 1: Comparison: Placebo/Docetaxel vs Aflibercept/Docetaxel; Test type: Superiority or Other; p = 0.0035, Stratified Log-Rank test; Stratified on ECOG Performance Status (0 vs 1 vs 2) and Prior Bevacizumab (yes vs no) according to IVRS; Stratified Hazard ratio = 0.819, 95% CI 2-sided [0.716 to 0.937] — Stratified on ECOG Performance Status (0 vs 1 vs 2) and Prior Bevacizumab (yes vs no) according to IVRS

3. Secondary Outcome: Overall Response (OR) Rate as Per Response Evaluation Criteria in Solid Tumours (RECIST) Criteria
Description: Participants with OR were those who had a confirmed complete response [CR] or a confirmed partial response [PR], based on RECIST criteria, in which
  * CR refected the disappearance of all tumor lesions (with no new tumors)
  * PR reflected a pre-defined decrease in tumor burden - a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  * OR was CR + PR The response rate was the percent of participants with a response.
  To determine a response, tumors were assessed by the investigators using Computerized Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans; and an observed response was confirmed by repeated imaging after 4 - 6 weeks.
Time Frame: Baseline to data cut-off (26 January 2011)
Population: Evaluable population: All ITT participants with measurable disease at study entry, and with at least one valid post baseline tumor evaluation, except if the participant died due to progressive disease or had documented (ie, radiological) progression before having any post-baseline tumor evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Number analyzed (Participants) | 406 | 404
percentage of participants
  Complete Response (CR) rate | 0.2 | 0.2
  Partial Response (PR) rate | 8.6 | 23.0
  Overall Response (OR) rate | 8.9 | 38.6

4. Secondary Outcome: Health Related Quality of Life (HRQL) Assessed by the Lung Cancer Symptom Scale (LCSS)
Description: HRQL assessments were performed by participants using a self-administered LCSS questionnaire. LCSS is a 9-item questionnaire, six measuring major symptoms for lung malignancies (appetite, fatigue, cough, dyspnea, hemoptysis and pain), and 3 summation items related to total symptomatic distress, activity status and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-mm lines. The LCSS total score was defined as the mean of the 9 items of the scale, each scored between 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline (prior to first dose), at cycles 2 and 4 and at the end of study therapy.
Population: ITT population with questionnaires evaluable for LCSS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Number analyzed (Participants) | 457 | 456
units on a scale
  Baseline (N=431, N=428) | 29.52 (17.03) | 31.54 (18.03)
  Cycle 2 (N=329, N=315) | 29.50 (16.72) | 30.54 (16.78)
  Cycle 4 (N=211, N=240) | 27.67 (16.24) | 29.61 (16.92)
  End of treatment (N=254, N=240) | 34.82 (18.34) | 36.07 (18.81)

5. Secondary Outcome: Health Related Quality of Life (HRQL) Assessed by the Average Symptom Burden Index (ASBI)
Description: HRQL assessments were performed by participants using a self-administered LCSS questionnaire. LCSS is a 9-item questionnaire, six measuring major symptoms for lung malignancies, and 3 summation items related to total symptomatic distress, activity status and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-mm lines. ABSI was the mean score for the six major lung cancer symptoms (appetite, fatigue, cough, dyspnea, hemoptysis and pain), each scored between 0 (for best outcome) to 100 (for worst outcome).
Time Frame: Baseline (prior to first dose), at cycles 2 and 4 and at the end of study therapy.
Population: ITT population with questionnaires evaluable for ABSI.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Number analyzed (Participants) | 457 | 456
units on a scale
  Baseline (N=429, N=429) | 26.17 (16.30) | 28.24 (16.91)
  Cycle 2 (N=327, N=316) | 26.23 (15.93) | 27.05 (15.92)
  Cycle 4 (N=211, N=241) | 24.52 (15.22) | 26.19 (16.38)
  End of treatment (N=253, N=239) | 30.73 (17.26) | 31.19 (18.12)

ADVERSE EVENTS:
Time Frame: From treatment initiation to October 21, 2011
Description: A death event was reported as an SAE if it occurred within 30 days from end of study treatment, or if it occurred more than 30 days after the end of study treatment, and was due to adverse event. Death due to disease progression, 30 days after the end of study treatment is part of the efficacy endpoints (OS and PFS), but not the safety endpoints.
Arm/Group | Placebo/Docetaxel | Aflibercept/Docetaxel
Serious Adverse Events (participants affected / at risk) | 159/453 | 218/452
Other Adverse Events (participants affected / at risk) | 388/453 | 402/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Docetaxel (N=453) | Aflibercept/Docetaxel (N=452)
Pneumonia (Infections and infestations) | 20 | 15
Urinary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 4
Neutropenic infection (Infections and infestations) | 11 | 11
Respiratory tract infection (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Neutropenic sepsis (Infections and infestations) | 3 | 10
Lung infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 2
Empyema (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1
Hepatitis c (Infections and infestations) | 2 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Lung abscess (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 21
Neutropenia (Blood and lymphatic system disorders) | 7 | 16
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 6
Mental status changes (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 3
Hypotonia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebral artery thrombosis (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Nausea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Periproctitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Scrotal ulcer (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 1 | 4
Asthenia (General disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 5
Oedema peripheral (General disorders) | 1 | 0
Disease progression (General disorders) | 12 | 33
Pain (General disorders) | 0 | 2
Death (General disorders) | 3 | 7
Injection site reaction (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 3
General physical health deterioration (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Docetaxel (N=453) | Aflibercept/Docetaxel (N=452)
Decreased appetite (Metabolism and nutrition disorders) | 93 | 122
Peripheral sensory neuropathy (Nervous system disorders) | 65 | 54
Headache (Nervous system disorders) | 27 | 59
Dysgeusia (Nervous system disorders) | 15 | 35
Paraesthesia (Nervous system disorders) | 27 | 20
Lacrimation increased (Eye disorders) | 18 | 41
Hypertension (Vascular disorders) | 23 | 95
Cough (Respiratory, thoracic and mediastinal disorders) | 94 | 108
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 89 | 85
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 90
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 | 83
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 23 | 24
Stomatitis (Gastrointestinal disorders) | 69 | 180
Diarrhoea (Gastrointestinal disorders) | 106 | 124
Nausea (Gastrointestinal disorders) | 92 | 79
Constipation (Gastrointestinal disorders) | 55 | 65
Vomiting (Gastrointestinal disorders) | 56 | 57
Abdominal pain (Gastrointestinal disorders) | 25 | 20
Dysphagia (Gastrointestinal disorders) | 6 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 148 | 133
Nail disorder (Skin and subcutaneous tissue disorders) | 33 | 42
Rash (Skin and subcutaneous tissue disorders) | 26 | 30
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 43
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 38
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 31
Bone pain (Musculoskeletal and connective tissue disorders) | 22 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 19
Proteinuria (Renal and urinary disorders) | 4 | 34
Fatigue (General disorders) | 130 | 142
Asthenia (General disorders) | 84 | 83
Pyrexia (General disorders) | 42 | 53
Oedema peripheral (General disorders) | 54 | 29
Non-cardiac chest pain (General disorders) | 29 | 32
Weight decreased (Investigations) | 35 | 110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 30 days in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed 90 days).